CLINICAL TRIAL: NCT05532189
Title: ACL Reconstruction With Bone Tendon Bone (BTB) Autograft With Versus Without Internal Brace - Clinical and Radiographic Outcomes
Brief Title: Anterior Cruciate Ligament (ACL) Reconstruction With Bone Tendon Bone Autograft With Versus Without Internal Bracing
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAU0966
Record Dates: First submitted 2022-09-04; First posted 2022-09-08 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: ACL Tear
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to the ACL reconstruction without internal bracing group (control) or to the ACL reconstruction with internal bracing (experimental).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACL reconstruction with internal brace augmentation (suture tape) (Experimental): This group will receive a standard ACL reconstruction using a BTB autograft with suture tape augmentation on the graft to strengthen it during the surgical procedure.
  Interventions: Procedure: ACL reconstruction with BTB autograft with internal brace augmentation (suture tape); Other: Standardized Rehabilitation Protocol
- ACL reconstruction without internal brace augmentation (Active Comparator): This group will only receive a standard ACL reconstruction using a BTB autograft. No suture tape will be added to the graft during the surgical procedure.
  Interventions: Procedure: ACL reconstruction with BTB autograft without internal brace augmentation (suture tape); Other: Standardized Rehabilitation Protocol

INTERVENTIONS:
Procedure: ACL reconstruction with BTB autograft with internal brace augmentation (suture tape) — The ACL will be reconstructed using a participant's own patella tendon (BTB autograft), and the graft will be fortified by suture tape during the surgery in order to strengthen it.
  Arms: ACL reconstruction with internal brace augmentation (suture tape)
Procedure: ACL reconstruction with BTB autograft without internal brace augmentation (suture tape) — The ACL will be reconstructed using a participant's own patella tendon (BTB autograft). The graft will not be fortified by suture tape in this group. It will be used as is without any modification.
  Arms: ACL reconstruction without internal brace augmentation
Other: Standardized Rehabilitation Protocol — Participants will undergo a standardized rehabilitation protocol with twice weekly physical therapy

SUMMARY:
There is no consensus regarding the best surgical management of primary ACL tears. Recent evidence suggests that internal brace augmentation may increase load failure and therefore stabilize the graft in-situ at the time of ACL reconstruction. This prospective randomized controlled trial aims to compare the time to return to activity, and participant reported outcomes in participants with bone-tendon-bone ACL reconstruction with and without (control) internal brace augmentation.

DETAILED DESCRIPTION:
Despite the wide variety of surgical approaches and grafts that can be used in an ACL reconstruction, graft failure and recurrent knee instability are nevertheless ubiquitous issues that have facilitated interest in ways to strengthen the graft at the time of surgery. While both animal and biomechanical models have strongly suggested improved graft strength and patient outcomes by utilizing suture tape augmentation in ACL reconstructions, there is scant clinical literature available to assess these extrapolations. A retrospective cohort study of 60 patients undergoing ACL reconstruction with a hamstring autograft or allograft (30 suture tape vs 30 no suture tape; mean age: 30), found shorter time to return to activity (9.2 months suture tape group vs 12.9 months no suture tape group; p=0.002), lower Western Ontario and McMaster University Osteoarthritis Indices (WOMAC) (2.2 suture tape group vs 6.2 no suture tape group; p=0.024), higher international knee documentation committee (IKDC) scores (87.6 suture tape group vs 73.2 no suture tape group; p=0.006), lower average pain on the national pain rating scale (NPRS) (0.6 suture tape group vs 1.66 no suture tape group; p=0.021) and no significant difference in range of motion in degrees (129 suture tape group vs 127 no suture tape group; p=0.46), knee injury and osteoarthritis outcome score (KOOS) (92.2 suture tape group vs 87.1 no suture tape group; p=0.68), or complications (13% suture tape vs 10% no suture tape; p>0.05) at 2 years follow up. A retrospective cohort study of 108 patients undergoing ACL reconstruction with a hamstring autograft with and without suture tape reinforcement (36 suture tape vs 72 no suture tape; mean age: 25), found a significantly higher Tegner activity score (7.1 suture tape group vs 6.4 no suture tape group; p=0.026) but otherwise no significant difference in time to preinjury activity level (11.9 mos suture tape group vs 11.6 no suture tape group; p=0.59), range of motion (degrees) (136 suture tape group vs 137 no suture tape group; p=0.44) , Lysholm knee score (95.6 suture tape group vs 94 no suture tape group; p=0.165), IKDC score (94.4 suture tape group vs 93.8 no suture tape group; p=0.44), or complications (6% suture tape group vs 5% no suture tape group; p>0.05) at 2 years follow up. A prospective cohort study of 50 ACL reconstructions with hamstring autograft with and without suture tape reinforcement (25 suture tape group vs 25 no suture tape group; mean age: 30), found a significant improvement in greater than 2 grades of Lachman testing from preoperative assessment compared to 6 months follow-up (68% suture tape group vs 32% no suture tape group; p=0.039) but no difference in Lysholm knee score at 6 months (87.0 suture tape group vs 87.0 no suture tape group; p=0.756). Moreover, none of the already-limited clinical data investigates the use of internal braces with bone-tendon-bone grafts, which are a popular choice for young adults and athletes. Furthermore, there are no current level 1 data on this subject. Therefore, this study aims to compare the time to return to pre- injury activity level, incidence of recurrent knee instability, and patient reported outcomes of patients treated with ACL reconstruction using bone-tendon-bone autograft with and without (control group) internal brace stabilization.

ELIGIBILITY:
Inclusion Criteria:

* patients 12 and older
* patients seen by the Columbia University Sports Medicine Service
* patients diagnosed with a first time ACL injury by clinical exam and MRI

Exclusion Criteria:

* previous knee surgery
* concurrent knee fracture or ligamentous injury on ipsilateral knee
* neuromuscular disorder involving lower limb
* inability/ unwillingness to adhere to protocol
* anesthesia contraindications
* lost to follow up

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-09 (Estimated); Primary Completion 2032-09 (Estimated); Study Completion 2032-09 (Estimated)

PRIMARY OUTCOMES:
Time to Return to Full Activity or Sports | Measured once per participant, depending on the time required to return to full activity (up to 10 years)
  Time from treatment initiation to full return to pre-injury activity levels in each group, expressed in weeks
Percentage of Participants with Recurrent Knee Instability | 2 weeks, 6 weeks, 3 months, 6 months, 1 year, 2 years, 5 years and 10 years
  Percentage of participants that experience recurrent instability after treatment starts at each time point
Change in Patient Reported Outcome Measurement Information System (PROMIS) Physical Function (PF) Computer Adaptive Test (CAT) at 2 weeks | Baseline and 2 weeks
  A computerized questionnaire ranging from 0 to 100 points that addresses how a participant's physical functional capacity has been impacted by their knee injury. A lower score indicates a better outcome.
Change in PROMIS PF CAT at 6 weeks | Baseline and 6 weeks
  A computerized questionnaire ranging from 0 to 100 points that addresses how a participant's physical functional capacity has been impacted by their knee injury. A lower score indicates a better outcome.
Change in PROMIS PF CAT at 3 months | Baseline and 3 months
  A computerized questionnaire ranging from 0 to 100 points that addresses how a participant's physical functional capacity has been impacted by their knee injury. A lower score indicates a better outcome.
Change in PROMIS PF CAT at 6 months | Baseline and 6 months
  A computerized questionnaire ranging from 0 to 100 points that addresses how a participant's physical functional capacity has been impacted by their knee injury. A lower score indicates a better outcome.
Change in PROMIS PF CAT at 1 year | Baseline and 1 year
  A computerized questionnaire ranging from 0 to 100 points that addresses how a participant's physical functional capacity has been impacted by their knee injury. A lower score indicates a better outcome.
Change in PROMIS PF CAT at 2 years | Baseline and 2 years
  A computerized questionnaire ranging from 0 to 100 points that addresses how a participant's physical functional capacity has been impacted by their knee injury. A lower score indicates a better outcome.
Change in PROMIS PF CAT at 5 years | Baseline and 5 years
  A computerized questionnaire ranging from 0 to 100 points that addresses how a participant's physical functional capacity has been impacted by their knee injury. A lower score indicates a better outcome.
Change in PROMIS PF CAT at 10 years | Baseline and 10 years
  A computerized questionnaire ranging from 0 to 100 points that addresses how a participant's physical functional capacity has been impacted by their knee injury. A lower score indicates a better outcome.
Change in PROMIS Pain Interference (PI) CAT at 2 weeks | Baseline and 2 weeks
  A computerized questionnaire ranging from 0 to 100 points that addresses how a participant's pain has been impacted by their knee injury. A lower score indicates a better outcome.
Change in PROMIS PI CAT at 6 weeks | Baseline and 6 weeks
  A computerized questionnaire ranging from 0 to 100 points that addresses how a participant's pain has been impacted by their knee injury. A lower score indicates a better outcome.
Change in PROMIS PI CAT at 3 months | Baseline and 3 months
  A computerized questionnaire ranging from 0 to 100 points that addresses how a participant's pain has been impacted by their knee injury. A lower score indicates a better outcome.
Change in PROMIS PI CAT at 6 months | Baseline and 6 months
  A computerized questionnaire ranging from 0 to 100 points that addresses how a participant's pain has been impacted by their knee injury. A lower score indicates a better outcome.
Change in PROMIS PI CAT at 1 year | Baseline and 1 year
  A computerized questionnaire ranging from 0 to 100 points that addresses how a participant's pain has been impacted by their knee injury. A lower score indicates a better outcome.
Change in PROMIS PI CAT at 2 years | Baseline and 2 years
  A computerized questionnaire ranging from 0 to 100 points that addresses how a participant's pain has been impacted by their knee injury. A lower score indicates a better outcome.
Change in PROMIS PI CAT at 5 years | Baseline and 5 years
  A computerized questionnaire ranging from 0 to 100 points that addresses how a participant's pain has been impacted by their knee injury. A lower score indicates a better outcome.
Change in PROMIS PI CAT at 10 years | Baseline and 10 years
  A computerized questionnaire ranging from 0 to 100 points that addresses how a participant's pain has been impacted by their knee injury. A lower score indicates a better outcome.
Change in PROMIS Depression CAT at 2 weeks | Baseline and 2 weeks
  A computerized questionnaire ranging from 0 to 100 points that addresses how a participant's quality of life has been impacted by their knee injury. A lower score indicates a better outcome.
Change in PROMIS Depression CAT at 6 weeks | Baseline and 6 weeks
  A computerized questionnaire ranging from 0 to 100 points that addresses how a participant's quality of life has been impacted by their knee injury. A lower score indicates a better outcome.
Change in PROMIS Depression CAT at 3 months | Baseline and 3 months
  A computerized questionnaire ranging from 0 to 100 points that addresses how a participant's quality of life has been impacted by their knee injury. A lower score indicates a better outcome.
Change in PROMIS Depression CAT at 6 months | Baseline and 6 months
  A computerized questionnaire ranging from 0 to 100 points that addresses how a participant's quality of life has been impacted by their knee injury. A lower score indicates a better outcome.
Change in PROMIS Depression CAT at 1 year | Baseline and 1 year
  A computerized questionnaire ranging from 0 to 100 points that addresses how a participant's quality of life has been impacted by their knee injury. A lower score indicates a better outcome.
Change in PROMIS Depression CAT at 2 years | Baseline and 2 years
  A computerized questionnaire ranging from 0 to 100 points that addresses how a participant's quality of life has been impacted by their knee injury. A lower score indicates a better outcome.
Change in PROMIS Depression CAT at 5 years | Baseline and 5 years
  A computerized questionnaire ranging from 0 to 100 points that addresses how a participant's quality of life has been impacted by their knee injury. A lower score indicates a better outcome.
Change in PROMIS Depression CAT at 10 years | Baseline and 10 years
  A computerized questionnaire ranging from 0 to 100 points that addresses how a participant's quality of life has been impacted by their knee injury. A lower score indicates a better outcome.

SECONDARY OUTCOMES:
Change in Western Ontario and McMaster Universities Arthritis Index (WOMAC) Score at 2 weeks | Baseline and 2 weeks
  The WOMAC questionnaire has subscores for pain (0-20), stiffness (0-8), and physical function (0-68), which address the impact of an injury on a participant's life. A lower total score (sum of subscores) indicates a better outcome.
Change in Western Ontario and McMaster Universities Arthritis Index (WOMAC) Score at 6 weeks | Baseline and 6 weeks
  The WOMAC questionnaire has subscores for pain (0-20), stiffness (0-8), and physical function (0-68), which address the impact of an injury on a participant's life. A lower total score (sum of subscores) indicates a better outcome.
Change in Western Ontario and McMaster Universities Arthritis Index (WOMAC) Score at 3 months | Baseline and 3 months
  The WOMAC questionnaire has subscores for pain (0-20), stiffness (0-8), and physical function (0-68), which address the impact of an injury on a participant's life. A lower total score (sum of subscores) indicates a better outcome.
Change in Western Ontario and McMaster Universities Arthritis Index (WOMAC) Score at 6 months | Baseline and 6 months
  The WOMAC questionnaire has subscores for pain (0-20), stiffness (0-8), and physical function (0-68), which address the impact of an injury on a participant's life. A lower total score (sum of subscores) indicates a better outcome.
Change in Western Ontario and McMaster Universities Arthritis Index (WOMAC) Score at 1 year | Baseline and 1 year
  The WOMAC questionnaire has subscores for pain (0-20), stiffness (0-8), and physical function (0-68), which address the impact of an injury on a participant's life. A lower total score (sum of subscores) indicates a better outcome.
Change in Western Ontario and McMaster Universities Arthritis Index (WOMAC) Score at 2 years | Baseline and 2 years
  The WOMAC questionnaire has subscores for pain (0-20), stiffness (0-8), and physical function (0-68), which address the impact of an injury on a participant's life. A lower total score (sum of subscores) indicates a better outcome.
Change in Western Ontario and McMaster Universities Arthritis Index (WOMAC) Score at 5 years | Baseline and 5 years
  The WOMAC questionnaire has subscores for pain (0-20), stiffness (0-8), and physical function (0-68), which address the impact of an injury on a participant's life. A lower total score (sum of subscores) indicates a better outcome.
Change in Western Ontario and McMaster Universities Arthritis Index (WOMAC) Score at 10 years | Baseline and 10 years
  The WOMAC questionnaire has subscores for pain (0-20), stiffness (0-8), and physical function (0-68), which address the impact of an injury on a participant's life. A lower total score (sum of subscores) indicates a better outcome.
Change in International Knee Documentation Committee (IKDC) Score at 2 weeks | Baseline and 2 weeks
  The IKDC questionnaire is scored from 0 (worse outcome)-100 (better outcome) and addresses knee symptoms, function, and physical activity.
Change in International Knee Documentation Committee (IKDC) Score at 6 weeks | Baseline and 6 weeks
  The IKDC questionnaire is scored from 0 (worse outcome)-100 (better outcome) and addresses knee symptoms, function, and physical activity.
Change in International Knee Documentation Committee (IKDC) Score at 3 months | Baseline and 3 months
  The IKDC questionnaire is scored from 0 (worse outcome)-100 (better outcome) and addresses knee symptoms, function, and physical activity.
Change in International Knee Documentation Committee (IKDC) Score at 6 months | Baseline and 6 months
  The IKDC questionnaire is scored from 0 (worse outcome)-100 (better outcome) and addresses knee symptoms, function, and physical activity.
Change in International Knee Documentation Committee (IKDC) Score at 1 year | Baseline and 1 year
  The IKDC questionnaire is scored from 0 (worse outcome)-100 (better outcome) and addresses knee symptoms, function, and physical activity.
Change in International Knee Documentation Committee (IKDC) Score at 2 years | Baseline and 2 years
  The IKDC questionnaire is scored from 0 (worse outcome)-100 (better outcome) and addresses knee symptoms, function, and physical activity.
Change in International Knee Documentation Committee (IKDC) Score at 5 years | Baseline and 5 years
  The IKDC questionnaire is scored from 0 (worse outcome)-100 (better outcome) and addresses knee symptoms, function, and physical activity.
Change in International Knee Documentation Committee (IKDC) Score at 10 years | Baseline and 10 years
  The IKDC questionnaire is scored from 0 (worse outcome)-100 (better outcome) and addresses knee symptoms, function, and physical activity.
Change in numeric pain rating scale (NPRS) Score at 2 weeks | Baseline and 2 weeks
  The NPRS is a questionnaire on a visual analog scale of 0 to 10 that a participant rates based on how bad their pain is (0 = no pain; 10 = maximum pain)
Change in numeric pain rating scale (NPRS) Score at 6 weeks | Baseline and 6 weeks
  The NPRS is a questionnaire on a visual analog scale of 0 to 10 that a participant rates based on how bad their pain is (0 = no pain; 10 = maximum pain)
Change in numeric pain rating scale (NPRS) Score at 3 months | Baseline and 3 months
  The NPRS is a questionnaire on a visual analog scale of 0 to 10 that a participant rates based on how bad their pain is (0 = no pain; 10 = maximum pain)
Change in numeric pain rating scale (NPRS) Score at 6 months | Baseline and 6 months
  The NPRS is a questionnaire on a visual analog scale of 0 to 10 that a participant rates based on how bad their pain is (0 = no pain; 10 = maximum pain)
Change in numeric pain rating scale (NPRS) Score at 1 year | Baseline and 1 year
  The NPRS is a questionnaire on a visual analog scale of 0 to 10 that a participant rates based on how bad their pain is (0 = no pain; 10 = maximum pain)
Change in numeric pain rating scale (NPRS) Score at 2 years | Baseline and 2 years
  The NPRS is a questionnaire on a visual analog scale of 0 to 10 that a participant rates based on how bad their pain is (0 = no pain; 10 = maximum pain)
Change in numeric pain rating scale (NPRS) Score at 5 years | Baseline and 5 years
  The NPRS is a questionnaire on a visual analog scale of 0 to 10 that a participant rates based on how bad their pain is (0 = no pain; 10 = maximum pain)
Change in numeric pain rating scale (NPRS) Score at 10 years | Baseline and 10 years
  The NPRS is a questionnaire on a visual analog scale of 0 to 10 that a participant rates based on how bad their pain is (0 = no pain; 10 = maximum pain)
Change in Knee Injury and Osteoarthritis Outcome Score (KOOS) at 2 weeks | Baseline and 2 weeks
  The KOOS score is a questionnaire regarding the severity of participants' knee symptoms, which is scored from 0 to 100 (100 representing no severity; 0 representing maximum severity )
Change in Knee Injury and Osteoarthritis Outcome Score (KOOS) at 6 weeks | Baseline and 6 weeks
  The KOOS score is a questionnaire regarding the severity of participants' knee symptoms, which is scored from 0 to 100 (100 representing no severity; 0 representing maximum severity )
Change in Knee Injury and Osteoarthritis Outcome Score (KOOS) at 3 months | Baseline and 3 months
  The KOOS score is a questionnaire regarding the severity of participants' knee symptoms, which is scored from 0 to 100 (100 representing no severity; 0 representing maximum severity )
Change in Knee Injury and Osteoarthritis Outcome Score (KOOS) at 6 months | Baseline and 6 months
  The KOOS score is a questionnaire regarding the severity of participants' knee symptoms, which is scored from 0 to 100 (100 representing no severity; 0 representing maximum severity )
Change in Knee Injury and Osteoarthritis Outcome Score (KOOS) at 1 year | Baseline and 1 year
  The KOOS score is a questionnaire regarding the severity of participants' knee symptoms, which is scored from 0 to 100 (100 representing no severity; 0 representing maximum severity )
Change in Knee Injury and Osteoarthritis Outcome Score (KOOS) at 2 years | Baseline and 2 years
  The KOOS score is a questionnaire regarding the severity of participants' knee symptoms, which is scored from 0 to 100 (100 representing no severity; 0 representing maximum severity )
Change in Knee Injury and Osteoarthritis Outcome Score (KOOS) at 5 years | Baseline and 5 years
  The KOOS score is a questionnaire regarding the severity of participants' knee symptoms, which is scored from 0 to 100 (100 representing no severity; 0 representing maximum severity )
Change in Knee Injury and Osteoarthritis Outcome Score (KOOS) at 10 years | Baseline and 10 years
  The KOOS score is a questionnaire regarding the severity of participants' knee symptoms, which is scored from 0 to 100 (100 representing no severity; 0 representing maximum severity )
Change in Tegner activity scale (TAS) Score at 2 weeks | Baseline and 2 weeks
  TAS is a one-item questionnaire assessing the activity level of patients on a scale of 0-10, with 0 representing disability and 10 representing the level of a professional athlete.
Change in Tegner activity scale (TAS) Score at 6 weeks | Baseline and 6 weeks
  TAS is a one-item questionnaire assessing the activity level of patients on a scale of 0-10, with 0 representing disability and 10 representing the level of a professional athlete.
Change in Tegner activity scale (TAS) Score at 3 months | Baseline and 3 months
  TAS is a one-item questionnaire assessing the activity level of patients on a scale of 0-10, with 0 representing disability and 10 representing the level of a professional athlete.
Change in Tegner activity scale (TAS) Score at 6 months | Baseline and 6 months
  TAS is a one-item questionnaire assessing the activity level of patients on a scale of 0-10, with 0 representing disability and 10 representing the level of a professional athlete.
Change in Tegner activity scale (TAS) Score at 1 year | Baseline and 1 year
  TAS is a one-item questionnaire assessing the activity level of patients on a scale of 0-10, with 0 representing disability and 10 representing the level of a professional athlete.
Change in Tegner activity scale (TAS) Score at 2 years | Baseline and 2 years
  TAS is a one-item questionnaire assessing the activity level of patients on a scale of 0-10, with 0 representing disability and 10 representing the level of a professional athlete.
Change in Tegner activity scale (TAS) Score at 5 years | Baseline and 5 years
  TAS is a one-item questionnaire assessing the activity level of patients on a scale of 0-10, with 0 representing disability and 10 representing the level of a professional athlete.
Change in Tegner activity scale (TAS) Score at 10 years | Baseline and 10 years
  TAS is a one-item questionnaire assessing the activity level of patients on a scale of 0-10, with 0 representing disability and 10 representing the level of a professional athlete.
Change in Lysholm Score at 2 weeks | Baseline and 2 weeks
  Lysholm score is a questionnaire out of 100 points that addresses specific aspects of participant's knee symptoms, with 100 indicating little to no symptoms and 0 indicating severe symptoms.
Change in Lysholm Score at 6 weeks | Baseline and 6 weeks
  Lysholm score is a questionnaire out of 100 points that addresses specific aspects of participant's knee symptoms, with 100 indicating little to no symptoms and 0 indicating severe symptoms.
Change in Lysholm Score at 3 months | Baseline and 3 months
  Lysholm score is a questionnaire out of 100 points that addresses specific aspects of participant's knee symptoms, with 100 indicating little to no symptoms and 0 indicating severe symptoms.
Change in Lysholm Score at 6 months | Baseline and 6 months
  Lysholm score is a questionnaire out of 100 points that addresses specific aspects of participant's knee symptoms, with 100 indicating little to no symptoms and 0 indicating severe symptoms.
Change in Lysholm Score at 1 year | Baseline and 1 year
  Lysholm score is a questionnaire out of 100 points that addresses specific aspects of participant's knee symptoms, with 100 indicating little to no symptoms and 0 indicating severe symptoms.
Change in Lysholm Score at 2 years | Baseline and 2 years
  Lysholm score is a questionnaire out of 100 points that addresses specific aspects of participant's knee symptoms, with 100 indicating little to no symptoms and 0 indicating severe symptoms.
Change in Lysholm Score at 5 years | Baseline and 5 years
  Lysholm score is a questionnaire out of 100 points that addresses specific aspects of participant's knee symptoms, with 100 indicating little to no symptoms and 0 indicating severe symptoms.
Change in Lysholm Score at 10 years | Baseline and 10 years
  Lysholm score is a questionnaire out of 100 points that addresses specific aspects of participant's knee symptoms, with 100 indicating little to no symptoms and 0 indicating severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: David P Trofa, MD, Principal Investigator — Associate Professor of Orthopaedic Surgery
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mall NA, Chalmers PN, Moric M, Tanaka MJ, Cole BJ, Bach BR Jr, Paletta GA Jr. Incidence and trends of anterior cruciate ligament reconstruction in the United States. Am J Sports Med. 2014 Oct;42(10):2363-70. doi: 10.1177/0363546514542796. Epub 2014 Aug 1. PMID 25086064
- [Background] Cohen SB, Yucha DT, Ciccotti MC, Goldstein DT, Ciccotti MA, Ciccotti MG. Factors affecting patient selection of graft type in anterior cruciate ligament reconstruction. Arthroscopy. 2009 Sep;25(9):1006-10. doi: 10.1016/j.arthro.2009.02.010. PMID 19732639
- [Background] Spindler KP, Wright RW. Clinical practice. Anterior cruciate ligament tear. N Engl J Med. 2008 Nov 13;359(20):2135-42. doi: 10.1056/NEJMcp0804745. No abstract available. PMID 19005197
- [Background] Engebretsen L, Benum P, Fasting O, Molster A, Strand T. A prospective, randomized study of three surgical techniques for treatment of acute ruptures of the anterior cruciate ligament. Am J Sports Med. 1990 Nov-Dec;18(6):585-90. doi: 10.1177/036354659001800605. PMID 2285086
- [Background] Bowman EN, Limpisvasti O, Cole BJ, ElAttrache NS. Anterior Cruciate Ligament Reconstruction Graft Preference Most Dependent on Patient Age: A Survey of United States Surgeons. Arthroscopy. 2021 May;37(5):1559-1566. doi: 10.1016/j.arthro.2021.01.042. Epub 2021 Feb 1. PMID 33539983
- [Background] Bodendorfer BM, Michaelson EM, Shu HT, Apseloff NA, Spratt JD, Nolton EC, Argintar EH. Suture Augmented Versus Standard Anterior Cruciate Ligament Reconstruction: A Matched Comparative Analysis. Arthroscopy. 2019 Jul;35(7):2114-2122. doi: 10.1016/j.arthro.2019.01.054. Epub 2019 Jun 2. PMID 31167738
- [Background] Parkes CW, Leland DP, Levy BA, Stuart MJ, Camp CL, Saris DBF, Krych AJ. Hamstring Autograft Anterior Cruciate Ligament Reconstruction Using an All-Inside Technique With and Without Independent Suture Tape Reinforcement. Arthroscopy. 2021 Feb;37(2):609-616. doi: 10.1016/j.arthro.2020.09.002. Epub 2020 Nov 2. PMID 33144236
- [Background] Batty LM, Norsworthy CJ, Lash NJ, Wasiak J, Richmond AK, Feller JA. Synthetic devices for reconstructive surgery of the cruciate ligaments: a systematic review. Arthroscopy. 2015 May;31(5):957-68. doi: 10.1016/j.arthro.2014.11.032. Epub 2015 Jan 22. PMID 25620500
- [Background] Smith PA, Bley JA. Allograft Anterior Cruciate Ligament Reconstruction Utilizing Internal Brace Augmentation. Arthrosc Tech. 2016 Oct 10;5(5):e1143-e1147. doi: 10.1016/j.eats.2016.06.007. eCollection 2016 Oct. PMID 28224069
- [Background] E A Mackenzie C, Huntington LS, Tulloch S. Suture Tape Augmentation of Anterior Cruciate Ligament Reconstruction Increases Biomechanical Stability: A Scoping Review of Biomechanical, Animal, and Clinical Studies. Arthroscopy. 2022 Jun;38(6):2073-2089. doi: 10.1016/j.arthro.2021.12.036. Epub 2022 Jan 3. PMID 34990759